CLINICAL TRIAL: NCT05807282
Title: Interventions to Decrease Heat Stress Among Latinx Farmworkers in Idaho
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not funded
Sponsor: Boise State University (Other)
Responsible Party: Principal Investigator, Carly Hyland, Assistant Prfoessor, Boise State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BoiseSU
Record Dates: First submitted 2023-03-17; First posted 2023-04-11 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Environmental Exposure
Keywords: farmworker; heat exposure

STUDY DESIGN:
Intervention Model Description: 80 farmworkers identifying as Hispanic/Latinx will be randomized to one of two treatment arms: 1) individual- and workplace-level interventions to decrease the health impacts of occupational heat stress, or 2) control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 40 farmworkers will be randomized to receive the workplace- and individual-level interventions developed in collaboration with study partners (e.g., provision of hydration packs to participants). Participants will receive the intervention at the workplace and will be monitored for five weeks after the intervention to evaluate the efficacy in reducing perceived and physiological heat stress.
  Interventions: Other: Interventions to Decrease Heat Stress among Latinx Farmworkers in Idaho
- Control group (No Intervention): 40 farmworkers will be randomized to receive no intervention, and will continue their work as normal. These farmworkers will be monitored for the same period as the intervention group to assess perceived and physiological heat stress.

INTERVENTIONS:
Other: Interventions to Decrease Heat Stress among Latinx Farmworkers in Idaho — The interventions will be developed in collaboration with our study partners and will include increasing access to shade at the workplace, providing hydration packs to participants, and providing education regarding the signs and symptoms of occupational heat stress.
  Arms: Intervention group

SUMMARY:
The goal of this study is to collaborate with farmworker, community organizations, and labor contractors/employers to develop workplace- and individual-level interventions, and evaluate the efficacy of those interventions in decreasing physiological and perceived heat stress among Latinx farmworkers in Idaho.

DETAILED DESCRIPTION:
Occupational heat exposure presents one of the clearest acute and long-term health threats to farmworkers and will continue to worsen under climate change. Exposure to extreme heat can lead to Heat-Related Illnesses (HRI), a continuum of diseases that can range from mild symptoms (e.g., dizziness, fatigue, vomiting) to severe and life-threatening conditions including convulsions, coma, and even death. It is becoming increasingly urgent to identify effective strategies to prevent the health impacts of heat exposure among farmworkers as climate change increases the frequency, intensity, and duration of heat waves. The few studies that have examined this topic have identified some beneficial impacts of increasing access to cold water and shade at the workplace, however studies to date have been limited by their investigation of individual- and workplace- interventions in isolation and research teams that do not engage farmworkers and community-based organizations. Further, the studies that have been conducted have taken place primarily in states with regulations that prohibit work over a specific heat index, and it is important to examine the impacts of interventions to decrease heat stress in states without these regulations, such as Idaho. The aims of this study are to collaborate with farmworkers, farmworker employers, and community organizations to develop and evaluate the efficacy of multi-level interventions in mitigating physiological and perceived heat strain among Latinx farmworkers in Idaho. The investigators further aim to examine the efficacy of educational programs (e.g., training in identifying and preventing personal and occupational risk factors for heat stress) on knowledge, behaviors, and perceptions. Leveraging our existing and well-established relationships with multiple community partners, the investigators will disseminate the research findings and promote the implementation of health-protective heat interventions to farmworkers, farmworker employers, and stakeholders across Idaho and the Mountain West. This study was motivated by concerns voiced by participants in a previous study of Latinx farmworkers led by the current team of researchers and community organizations. Here, the investigators aim to respond directly to their stated concerns regarding occupational heat exposure.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Hispanic/Latinx, currently working in an agricultural field in Idaho

Exclusion Criteria:

* Under age 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-16 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Body temperature | Up to 10 weeks
  The investigators will use sensors to monitor participants' body temperature as a sign of physiological heat stress. The investigators will compare differences in physiological heat stress between the control and intervention groups.
Heart rate | Up to 10 weeks
  The investigators will use sensors to monitor participants' heart rate as a sign of physiological heat stress. The investigators will compare differences in physiological heat stress between the control and intervention groups.

SECONDARY OUTCOMES:
Perceived heat stress (questionnaire) | Up to 10 weeks
  The investigators will administer weekly questionnaires assessing participants' perceived heat stress (e.g., self-report of nausea, vomiting and fatigue). The investigators will assess 15 symptoms and compare differences in the number of symptoms reported between the control and intervention groups.

IPD SHARING:
Plan to Share IPD: No
In order to protect the confidentiality of this structurally marginalized population, data from this study will not be shared with outside investigators.